CLINICAL TRIAL: NCT05410236
Title: The Application of Three-dimensional Printing in Airway Anatomy and Bronchoscopy Education
Brief Title: 3D Printing in Airway Anatomy and Bronchoscopy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapy, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PL202008018V
Record Dates: First submitted 2022-02-25; First posted 2022-06-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Satisfaction, Personal
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimatal (Experimental): Learning anatomy with 3D bronchial tree model.
  Interventions: Other: 3D bronchial tree model
- Control group (No Intervention): Learning anatomy without 3D bronchial tree model.

INTERVENTIONS:
Other: 3D bronchial tree model — A detachable 3D printed bronchial tree model
  Arms: Experimatal

SUMMARY:
The main purpose of this study is to use 3D printing technology to make a human anatomical bronchial tree model, which is applied in medical education for medical students and students of the department of respiratory therapy. Most of the clinical teaching material is expansive and inaccessible. To promote accessibility of anatomy models and student learning effects in our school and hospital, we use the 3D printing technology to print bronchial tree model and apply it to anatomy and bronchoscopy education.

The present study expects some benefits that the use of printed bronchial trees for anatomy and bronchoscopy education. For example, it can reduce the cost of anatomy instruction, let students have their own anatomical model, and make the learning no longer limited to the anatomical classroom.

DETAILED DESCRIPTION:
Three-dimensional (3D) printing is a technology used for the rapid production of customized physical objects. Bronchoscopy is a well-established, relatively safe procedure for both diagnostic and therapeutic interventions for a variety of pulmonary diseases. In this study, to enhance the quality of airway anatomy education and bronchoscopy training, we used 3D printing to develop a 3D bronchial tree model as a high-fidelity simulator for bronchoscopy and demonstrated its validity. We designed a 3D bronchial tree model containing 12 detachable parts and 11 adapter rings.

ELIGIBILITY:
Inclusion Criteria:

* Student of Fu Jen Catholic University.

Exclusion Criteria:

* Refused to participate in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome.
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, MSc, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No